CLINICAL TRIAL: NCT00514995
Title: Sodium Oxybate in the Treatment of Binge Eating Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: Jazz Pharmaceuticals (Industry); University of Cincinnati (Other)
Responsible Party: Susan L. McElroy, MD / Professor, Lindner Center of HOPE and University of Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: McElroy
Record Dates: First submitted 2007-08-08; First posted 2007-08-10 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Sodium Oxybate

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Sodium Oxybate

INTERVENTIONS:
Drug: Sodium Oxybate — 4.5 g/night - 9 g/night, liquid taken twice per night

SUMMARY:
The purpose of this research study is to study the effectiveness, tolerability and safety of sodium oxybate in outpatients with binge eating disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patients will meet DSM-IV-TR criteria for BED for at least the last 6 months, determined by the Structured Clinical Interview for DSM-IV-TR (SCID) (72) and supported by the Eating Disorder Examination (EDE) (73). These criteria are as follows:

  * Recurrent episodes of binge eating. An episode of binge eating is characterized by both of the following:

    * eating, in discrete period of time (eg, within any two hour period), an amount of food that is definitely larger than most people would eat in a similar period of time under similar circumstances
    * a sense of lack of control over eating during the episode (eg, a feeling that one cannot stop eating or control what or how much one is eating)
  * The binge eating episodes are associated with at least three of the following:

    * eating much more rapidly than normal
    * eating until uncomfortably full
    * eating large amounts of food when not feeling physically hungry
    * eating alone because of being embarrassed by how much one is eating
    * feeling disgusted with oneself, depressed, or feeling very guilty after overeating
  * Marked distress regarding binge eating.
  * The binge eating occurs, on average, at least two days a week for six months.
  * Does not occur exclusively during the course of bulimia nervosa and anorexia nervosa.
* Men or women, from the ages of 21 through 65 years.
* Female subjects must either:

  * be incapable of pregnancy because of hysterectomy or tubal ligation.
  * if heterosexually active and capable of pregnancy, have been using an acceptable method of contraception (hormonal contraceptives, intrauterine device, spermicide and barrier or double barrier methods) for at least 1 month before study entry and agree to continue the use of one of these contraception methods for the duration of the study.
  * if sexually abstinent and capable of pregnancy, agree to continue abstinence or to use an acceptable method of birth control (either hormonal contraceptives, intrauterine device, spermicide and barrier or double barrier method) should sexual activity commence.

Exclusion Criteria:

* Have a current body mass index < 18kg/m2 or > 40kg/m2.
* Women who are pregnant or lactating and women of childbearing potential who are not taking adequate contraceptive measures. (All women of childbearing potential will have a negative pregnancy test before entering the study.)
* Subjects who are displaying current clinically significant depressive symptoms, defined as a Montgomery Asberg Depression Rating Scale (MADRS) (74) > 1324, or a major depressive episode by DSM-IV-TR criteria (1).
* Subjects who have a current or past history of clinically significant suicidality (as determined by psychiatric history, SCID interview, and MADRS suicide item #10) Subjects who have made > 1 lifetime suicide attempt and those with a MADRS suicide item score > 2 will be excluded from participation.
* Subjects who have a lifetime history of a DSM-IV-TR diagnosis of a substance abuse or dependence disorder, except for nicotine abuse or dependence (as determined by psychiatric history, SCID interview, and urine toxicology; see below).
* Subjects who have a lifetime history of a DSM-IV-TR psychotic disorder, bipolar disorder, or dementia.
* Subjects who have a history of a personality disorder (eg, schizotypal, borderline, or antisocial) which might interfere with assessment or compliance with study procedures.
* Clinically unstable medical disease, including cardiovascular, hepatic, renal, gastrointestinal, pulmonary, metabolic, endocrine or other systemic disease which could interfere with diagnosis, assessment, or treatment of binge eating disorder with sodium oxybate. Patients should be biochemically euthyroid prior to entering the study.
* History of obstructive sleep apnea (OBS) or receiving a high risk score for OBS on the Berlin Questionnaire (75).
* Subjects requiring treatment with any drug which might interact adversely with or obscure the action of the study medication (e.g. stimulants, sympathomimetics, antidepressants, carbonic anhydrase inhibitors, anti-obesity drugs, drugs with CNS depressant effects).
* Subjects who have received any psychoactive medication within one week prior to randomization.
* Subjects who have begun and/or are receiving formal psychotherapy (cognitive behavioral therapy, interpersonal therapy, or dietary behavioral therapy) for BED or weight loss within the past 3 months.
* Subjects previously enrolled in this study or have previously been treated with sodium oxybate.
* Subjects who have received an experimental drug or used an experimental device within 30 days.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the weekly frequency of binge-eating episodes (binge frequency). | 16 weeks

SECONDARY OUTCOMES:
Secondary outcome measures will include weekly frequency of binge days; body mass index; CGI-severity scores; YBOCS-BE modified for Binge Eating scores; Eating Inventory scores; and MADRS total scores. | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan L. McElroy, MD, Principal Investigator — University of Cincinnati
Locations (1):
- Lindner Center of HOPE, Mason, Ohio, United States

REFERENCES:
- [Result] McElroy SL, Guerdjikova AI, Winstanley EL, O'Melia AM, Mori N, Keck PE Jr, Hudson JI. Sodium oxybate in the treatment of binge eating disorder: an open-label, prospective study. Int J Eat Disord. 2011 Apr;44(3):262-8. doi: 10.1002/eat.20798. PMID 20209489